CLINICAL TRIAL: NCT07032779
Title: Effect of Simulation Application on Knowledge Level, Patient Safety Attitude and Self-Confidence Levels in Septic Shock Management
Brief Title: Effect of Simulation Application in Septic Shock Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NU-568
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Septic Shock
Keywords: simulation; education; nursing
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simulation (Experimental): After the septic shock scenario and preliminary preparations for the simulation to be used in the study are completed, the students in the intervention group will have the Tag Team Patient Safety Simulation application. The students in the simulation group will be divided into 2 groups and each group will have the Tag Team Patient Safety Simulation application with the same scenario. The students in the labeling group will be included in the scenario as the scenario progresses. It will start with 4 students at the beginning, but with labeling, 7-8 students in each group will take the role of the actors, and the other students will take the role of the audience. The simulation play will consist of a prologue, two acts, an intermission, an informational and an epilogue.
  Interventions: Other: simulation
- control (No Intervention): The students in the control group will not have the simulation application, and only the data collection forms will be filled out in the 2 specified time periods.

INTERVENTIONS:
Other: simulation — the students in the intervention group will have the Tag Team Patient Safety Simulation application. The students in the simulation group will be divided into 2 groups and each group will have the Tag Team Patient Safety Simulation application with the same scenario. The students in the labeling group will be included in the scenario as the scenario progresses. It will start with 4 students at the beginning, but with labeling, 7-8 students in each group will take the role of the actors, and the other students will take the role of the audience.
  Arms: simulation

SUMMARY:
This research will be conducted to determine the effect of the Tag Team Patient Safety Simulation application applied to second-year students of a university's Nursing Department on their knowledge level, patient safety attitudes and self-confidence levels.

DETAILED DESCRIPTION:
Introduction and Aim: Simulation education is a method that aims to provide students with artificial or virtual experience by providing them with a safe environment where real-life conditions are created. This research will be conducted to determine the effect of the Tag Team Patient Safety Simulation application applied to second-year students of a university's Nursing Department on their knowledge level, patient safety attitudes and self-confidence levels.

Methods: The research will be conducted in a quasi-experimental research design with a control group in a pre-test post-test design. The sample of the research will consist of students studying in the nursing department of a university and taking the Internal Medicine Nursing Course. Data will be collected in 2 time periods after theoretical information on the subject of septic shock is given, after the simulation application and at the end of the clinical application of the Internal Medicine Nursing course. After the septic shock scenario to be used in the research and the preliminary preparations for the simulation are completed, the students in the intervention group will be given the Tag Team Patient Safety Simulation application. No additional application will be made in the control group. Data were collected using the Personal Information Form, the Patient Safety Scale in Health Professional Education, the Student Satisfaction and Self-Confidence Scale in Learning, and the Septic Shock Knowledge Test.

Conclusions: As a result of the research, it is anticipated that the knowledge levels of students regarding patient care in shock will be increased, patient safety behaviors and self-confidence will be increased.Amasya University

ELIGIBILITY:
Inclusion Criteria:

* Students who are registered in the Internal Medicine Nursing course in the 2023-2024 academic year,
* Participated in the "Shock and Nursing Management" theoretical course in the Internal Medicine Nursing course,
* Completed the pre-test and post-tests in the study,
* Consent to the participate in the study

Exclusion Criteria:

* Students who did not participate in the theoretical and simulation application stages of the study,
* Did not consent to participate in the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Patient Safety in Education of Health Professionals Scale | 4 week
  Patient Safety in Education of Health Professionals Scale (SPEHGÖ): The Patient Safety in Education of Health Professionals Scale (SPEGHÖ); The scale; It has been reported as valid and reliable for the Turkish society with its original structure consisting of two main dimensions, 6 sub-dimensions, and 23 items. The scale; is a two-level measurement tool and consists of two main dimensions as "Class" and "Clinical environment". The six sub-dimensions in both main dimensions are; working as a team with other healthcare professionals (6 items), effective communication (3 items), management of security risks (3 items), understanding human and environmental factors (3 items), recognizing, intervening and revealing unexpected events and near-errors (4 items), safety culture (4 items). The increase in the total score average for the main and sub-dimensions indicates that the knowledge and competence regarding patient safety has increased
Student Satisfaction and Self-Confidence in Learning Scale | 4 week
  Student Satisfaction and Self-Confidence in Learning Scale: The validity and reliability study of the Student Satisfaction and Self-Confidence in Learning Scale in Turkish was conducted by Ünver et al. The total number of items was reduced to 12 during the adaptation of the scale to Turkish. The scale consists of the subheadings "Satisfaction with Current Learning" (5 items) and "Self-Confidence in Learning" (7 items). The sum of the sub-dimensions of the scale does not give the total score. As the total score obtained from the scale increases, student satisfaction and self-confidence in learning also increase
Septic Shock Knowledge Test | 4 week
  Septic Shock Knowledge Test: The knowledge test will consist of 15 questions regarding septic shock physiology, symptoms and treatment. The questions in the knowledge test will be sent to 5 experts and content validity will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- AmasyaU, Amasya, Turkey (Türkiye)